CLINICAL TRIAL: NCT06816329
Title: Tracking the Dynamic Trajectory of Behavioral, Physiological, and Neurobiological Stress Responses in Female Adolescents at High and Low Familial Risk for Depression
Brief Title: Stress Dynamics and Familial Risk for Depression in Female Adolescents
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mclean Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Emily L. Belleau, Assistant Professor, Mclean Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: R01MH137441 (NIH)
Record Dates: First submitted 2025-01-28; First posted 2025-02-10 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Major Depressive Disorder
Keywords: stress; depression; adolescents; neuroimaging; familial risk
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Intervention Model Description: Case-Control Design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Computer Task Manipulation (Experimental): Participants will complete computer tasks while undergoing an fMRI brain scan.
  Interventions: Behavioral: Computer Task Manipulation

INTERVENTIONS:
Behavioral: Computer Task Manipulation — Participants will complete computer tasks.

SUMMARY:
Stress and a parental history of major depressive disorder (MDD) are among the strongest risk factors for future development of MDD. Studies have shown that having a parental history of MDD may be associated with behavioral, psychophysiological, and hormonal responses to stress that are associated with poorer stress coping. . Adolescence is a vulnerable developmental window linked to increased MDD risk, especially for females, as rates of MDD surge relative to males. Despite the central role of stress in MDD onset, little is known about the brain mechanisms underlying stress responses in susceptible female adolescents at high familial risk for MDD. Also, it is unclear how stress-related brain network alterations may relate to "real-world" maladaptive stress responses and whether these stress-related brain network changes are predictive of future depression onset. We will fulfill these research gaps by combining neuroimaging with intensive longitudinal tracking of depressive symptomology as well as behavioral and physiological responses to "real world" stress using smartphone and smartwatch technology. Elucidating these neural mechanisms may aid in the discovery of MDD biomarkers that could identify youth at greatest risk for future MDD development and lead to earlier intervention efforts.

DETAILED DESCRIPTION:
Participants in this research study will include female adolescent between the age of 13 to 15, who may or may not have a parental history of depression. About 148 adolescents will take part in this study along with a biological parent/parent(s) over the next five years.

The study will include five sessions over the span of 18-months, including:

* A clinical diagnostic interview as well as filling out a series of questionnaires and assessments. This can be done virtually over Zoom or in-person.
* The second session will include a functional magnetic resonance imaging (fMRI) brain scan to be conducted at the McLean Hospital Imaging Center. Participants will be asked to respond to surveys on their cell phone in the two-weeks following the fMRI brain scan. Participants will also be given and asked to wear a smartwatch that tracks their heart rate, activity level, and sleep patterns for two-weeks.
* The third session will include a diagnostic interview, assessments, and questionnaires to be completed six-months after the fMRI brain scan. Participants will be asked to complete surveys on their cell phone during the two-weeks following this six month follow-up session. Participants will also be given and asked to wear a smartwatch that tracks their heart rate, activity level, and sleep patterns for two-weeks.
* The fourth session will include a diagnostic interview, assessments, and questionnaires to be completed 12-months after the fMRI brain scan. Participants will be asked to complete surveys on their cell phone during the two-weeks following this 12-month follow-up session. Participants will also be given and asked to wear a smartwatch that tracks their heart rate, activity level, and sleep patterns for two-weeks.
* The fifth session will include a diagnostic interview, assessments, and questionnaires to be completed 18-months after the fMRI brain scan. Participants will be asked to complete surveys on their cell phone during the two-weeks following this 18-month follow-up session. Participants will also be given and asked to wear a smartwatch that tracks their heart rate, activity level, and sleep patterns for two-weeks.

ELIGIBILITY:
Inclusion Criteria: General Inclusion Criteria for all Adolescent Cohorts:

* Female sex assigned at birth
* Ages 13-15
* English as first language or English Fluency
* Right-handed
* Have a personal cell phone to complete the ecological momentary assessments
* Ability to give signed, informed consent/assent either written or electronic (via RedCap eConsent)
* Normal or corrected to normal vision and hearing

Additional Inclusion Criteria for Female Adolescents with a Parental History of MDD, high-risk group:

• A biological parent meeting DSM-5 criteria for at least one past/current major depressive episode

Exclusion Criteria: General Exclusion Criteria for all Adolescent Cohorts:

• Presence of any contraindication for MRI:

* Cardiac pacemakers
* Metal clips on blood vessels (also called stents)
* Artificial heart valve, artificial arms, hands, legs, etc.
* Brain stimulator devices
* Implanted drug pumps
* Ear or eye implants
* Known metal fragments in eyes
* Exposure to metal filings or shrapnel (sheet metal workers, welders, and others)
* Other metallic surgical hardware in vital area
* Certain tattoos with metallic ink
* Certain intrauterine devices (IUDs) containing metal
* Any other metallic objects that are deemed a contraindication to MRI that cannot be removed
* Certain transdermal (skin) patches such as:

NicoDerm (nicotine for tobacco dependence) Transderm Scop (scopolamine for motion sickness) Ortho Evra (birth control)

* Presence of medical or neurological illness that could impact fMRI measures of cerebral blood flow (e.g., head injury resulting in loss of consciousness greater than 5 minutes, seizure, tic disorder, serious/unstable cardiac, hepatic, renal, respiratory, endocrine, neurologic or hematologic illnesses)
* Clinical/Laboratory Evidence of Hypothyroidism or Hyperthyroidism
* Use of hormonal replacement therapy, anabolic steroids
* Lifetime history of electroconvulsive therapy
* Current tobacco product use
* Lifetime use of any psychotropic medication
* Clinically significant levels of depressive symptoms according to the Children's Depression Rating Scale-Revised (T Score > 54, Poznanski et al., 1996)
* Diagnosis of a neurodevelopmental disorder (e.g., Autism Spectrum Disorder, Learning Disorder w/ impairment in reading) that would interfere with study tasks (e.g., understanding and completing lengthy battery of questionnaires, ability to complete fMRI scan session and tasks without moving)

Additional Exclusion Criteria for Female Adolescents with a Parental History of MDD, high-risk group:

• Lifetime or current Diagnostic and Statistical Manual (DSM)-5 diagnoses of MDD, persistent depressive disorder, schizophrenia spectrum or other psychotic disorder, bipolar disorder, substance/alcohol use disorder, eating disorders, and posttraumatic stress disorder

Additional Exclusion Criteria for Female Adolescents without a Parental History of MDD, low-risk group:

* Any past or current Diagnostic and Statistical Manual (DSM)-5 psychiatric or substance/alcohol use disorder
* First-degree relative history of any psychiatric disorder

Ages: 13 Years to 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Only female.
Enrollment: 148 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2030-03-31 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
Time Spent in Default Mode-Frontoparietal Network Coactivation Pattern (CAP) | Throughout a 1.75 hour MRI scan collected during the middle of a 3.5 hour 2nd study session
  Time Spent in Default Mode-Frontoparietal Network Coactivation Pattern (CAP). An fMRI variable. (the number of volumes spent in this CAP).
Persistence in default mode network-frontoparietal network co-activation pattern | Throughout a 1.75 hour MRI scan collected during the middle of a 3.5 hour 2nd study session
  Persistence in default mode network-frontoparietal network CAP. An fMRI measure. (the average number of consecutive volumes spent in this CAP)
Depressive Symptoms | Collected at baseline, the beginning of a 1.75 hour MRI, and at 6-, 12-, and 18-month follow-ups
  The total score on the Mood and Feelings Questionnaire [Min Score: 0, Max Score: 66, higher scores mean more severe depressive symptoms)

SECONDARY OUTCOMES:
Cortisol | Collected throughout a 3.5 hour second study session that involves a 1.75 hour MRI conducted at the middle of the session
  Saliva rating to be collected throughout the fMRI brain scan
Stress Ratings | Collected during a two-week period immediately after the 2nd study session (i.e., the MRI session), and then in the two-weeks immediately after the 6-, 12-, and 18-month follow-up sessions, respectively
  Stress ratings (0-100 sliding bar scale) collected via smartphone.
Average heart rate (beats per minute) | Collected during a two-week period immediately after the 2nd study session (i.e., the MRI session), and then in the two-weeks immediately after the 6-, 12-, and 18-month follow-up sessions, respectively
  compute average heart rate through smartwatch technology
heart rate variability | Collected during a two-week period immediately after the 2nd study session (i.e., the MRI session), and then in the two-weeks immediately after the 6-, 12-, and 18-month follow-up sessions, respectively
  heart rate variability expressed as the root mean square of successive differences (RMSSD)
Sleep duration | Collected during a two-week period immediately after the 2nd study session (i.e., the MRI session), and then in the two-weeks immediately after the 6-, 12-, and 18-month follow-up sessions, respectively
  sleep duration computed as the difference in minutes between sleep onset and sleep offset

CONTACTS AND LOCATIONS:
Overall Officials: Emily Belleau, Ph.D., Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Demographic, clinical, neuroimaging, psychophysiological, ecological momentary assessment, and smartwatch data will be preserved to enable sharing via NDA data of sufficient quality to validate and replicate research findings described in the Aims. NIMH requires data measured from human subjects to be shared using the NDA. All data will be deposited to NDA starting 12 months after the award begins and will be deposited every six months thereafter following the usual NDA data submission dates. Data will be findable for the research community through the NDA Collection that will be established when this application is funded. For all publications, an NDA study will be created. Each of those studies are assigned a digital object identifier (DOI). This data DOI will be referenced in the publication to allow the research community easy access to the exact data used in the publication. The research community will have access to data when the award ends.
Supporting Information: Analytic Code
Time Frame: The research community will have access to data when the award ends. NDA will make decisions about how long to preserve the data, but that data archive has not deleted any deposited data up to now.
Access Criteria: To request access of the data, researchers will use the standard processes at NDA, and the NDA Data Access Committee will decide which requests to grant. The standard NDA data access process allows access for one year and is renewable